CLINICAL TRIAL: NCT00049920
Title: The ARIC Neurocognitive Longitudinal Study
Brief Title: The ARIC MRI Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Thomas H. Mosley/Principal Investigator, University of Mississippi Medical center
Other Study IDs: 1194; R01HL070825 (NIH)
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-10

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Disorders; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To perform a follow-up study of cerebrovascular disease in the Atherosclerosis Risk in Communities (ARIC) magnetic resonance imaging subcohort.

DETAILED DESCRIPTION:
BACKGROUND:

Although the clinical manifestations of cerebrovascular disease (CVD) typically appear acutely, the deleterious effects of CVD on brain structure and function likely begin in a presymptomatic fashion at a younger age than clinical strokes. In an effort to characterize the prevalence, risk factors, and cognitive correlates of subclinical CVD, the Atherosclerosis Risk in Communities (ARIC) Study funded by the National Heart, Lung, and Blood Institute performed cerebral magnetic resonance imaging (MRI) and cognitive assessments on a large, bi-racial sample of middle-aged and young-elderly adults. Results from the ARIC MRI baseline study revealed a remarkably high prevalence of subclinical CVD including silent cerebral infarctions, white matter hyperintensities, and brain atrophy. Moreover, these subclinical abnormalities were found to be associated with reduced cognitive functioning and with clinical CVD outcomes such as incident stroke. Surprisingly little is known about risk factors related to the incidence or progression of subclinical CVD or how progression of these markers may relate to clinical outcomes such as stroke or neurocognitive decline.

DESIGN NARRATIVE:

This is a follow-up study of the ARIC MRI cohort, with repeated semiquantitative MR imaging and cognitive assessments. The study will also take advantage of recent advances in MR imaging and obtain volumetric measurements of selected brain regions and expand upon the baseline cognitive assessment to further characterize neurocognitive functioning. The longitudinal design of the proposed study will fill salient gaps in current understanding of subclinical CVD. Moreover, conducting this study within ARIC takes advantage of ARIC's baseline MRI data, unique African American population, and extensive vascular risk factor data (including new genetic and biochemical factors as well as subclinical markers of both large and small vessel disease), making an efficient study to provide new insights into the incidence, progression, and outcomes associated with subclinical CVD.

ELIGIBILITY:
Participated in the baseline ARIC MRI study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the ARIC Neurocognitive Longitudinal Study were recruited for a follow-up brain MR scan and cognitive testing from the subset of the (parent) ARIC cohort that had an initial MR scan at the third (Visit 3) ARIC examination. Participants included black and white men and women.
Sampling Method: Non-Probability Sample
Enrollment: 1134 (Actual)
Dates: Start 2002-09; Primary Completion 2006-05 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Mosley, PhD, Principal Investigator — University of Mississippi Medical Center

REFERENCES:
- [Background] Knopman DS, Mosley TH, Catellier DJ, Sharrett AR; Atherosclerosis Risk in Communities (ARIC) Study. Cardiovascular risk factors and cerebral atrophy in a middle-aged cohort. Neurology. 2005 Sep 27;65(6):876-81. doi: 10.1212/01.wnl.0000176074.09733.a8. PMID 16186527